CLINICAL TRIAL: NCT03527160
Title: Assessment of Urinary Neutrophil Gelatinase-Associated Lipocalin to Predict Acute Kidney Injury in Children Research Multiple Nephrotoxic Medications
Brief Title: Assessment of Urinary NGAL to Predict AKI in Children Receiving Multiple Nephrotoxic Medications
Acronym: NINJA NGAL
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: BioPorto Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CIN001 - NINJA NGAL
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Kidney Injury; Nephrotoxicity
Keywords: AKI; NGAL
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nephrotoxic medication (NTMx) exposure is one of the most commonly cited causes of acute kidney injury (AKI) in hospitalized children, and is the primary cause of AKI in 16% of cases. Through initial work at Cincinnati Children's Medical Center, NTMx exposure was found to be potentially modifiable and the associated AKI is an avoidable adverse safety event. Currently, only serum Creatinine monitoring is available to monitor for NTMx-associated AKI. The hypotheses of this NINJA NGAL study are that (1) urine NGAL is highly sensitive to detect NTMx-associated AKI, and (2) Bedside test of urine from high risk NTMx-exposed patients are adequate and reliable compared to urine NGAL measured from the clinical platform.

ELIGIBILITY:
Inclusion Criteria:

* Receiving 3 or more nephrotoxic medications on the same day OR
* Receiving 3 or more days of an intravenous aminoglycoside or vancomycin

Exclusion Criteria:

* Currently being treated for a urinary tract infection
* Presence of an acute kidney injury prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients in non-ICU settings at participating pediatric institutions
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's of Alabama, Birmingham, Alabama
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NINJA: Inpatients exposed to nephrotoxic medications
Period: Overall Study
Arm/Group | NINJA
Started | 134
Completed | 113
Not Completed | 21
Not completed — No urine collected | 13
Not completed — No clinical serum creatinine collected | 6
Not completed — Did not meet inclusion | 2

BASELINE CHARACTERISTICS:
Population: Participants separated into these two groups during the analysis, depending on whether they developed AKI per KDIGO serum creatinine guidelines during the course of their participation in the study.
Groups:
- Any AKI: Patients developed AKI during study
- No AKI: Patients did not develop AKI over the course of the study
- Total: Total of all reporting groups
Arm/Group | Any AKI | No AKI | Total
Number analyzed (Participants) | 27 | 86 | 113
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.2 [12.1 to 19.1] | 12.0 [5.9 to 18.0] | 13.2 [6.7 to 18.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 45 | 52
  Male | 20 | 41 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 27 | 83 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 12 | 15
  White | 24 | 66 | 90
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 5 | 5
Weight [Median (Inter-Quartile Range); unit: kilograms] | 47.1 [32.5 to 66.3] | 39.9 [18.0 to 53.0] | 42.3 [21.0 to 56.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Nephrotoxic Medication Associated AKI Detected by Urinary NGAL
Description: AKI, defined as a 50% rise in serum Creatinine over baseline or a 0.3 mg/dL rise within 48 hours, will be first detected by a rise in Urinary NGAL
Time Frame: 9 Days
Measure: Count of Participants; unit: Participants
Groups:
- Any AKI: Patients developed Nephrotoxic Medication Associated AKI during study
- No AKI: Patients did not develop Nephrotoxic Medication Associated AKI over the course of the study
Arm/Group | Any AKI | No AKI
Number analyzed (Participants) | 27 | 86
Participants
  NGAL >= 150 ng/mL | 3 | 6
  NGAL < 150 ng/mL | 24 | 80

2. Secondary Outcome: Point of Care NGAL Reliability Compared to Clinical Urinary NGAL
Description: A POC urinary NGAL will be determined from a colorimetric assay that determines risk of AKI, which will later be compared to NGAL values from the clinical assay
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Groups:
- NGAL >= 150 ng/mL: Participants who had an elevated point of care urine NGAL
- NGAL<150 ng/mL: Point of care urine NGAL less than 150 ng/mL
Arm/Group | NGAL >= 150 ng/mL | NGAL<150 ng/mL
Number analyzed (Participants) | 51 | 62
Participants
  AKI | 10 | 16
  No AKI | 41 | 46

ADVERSE EVENTS:
Time Frame: Maximum of 9 days of exposure
Description: Adverse events were defined as any sign, symptoms, illness, clinically significant abnormal laboratory value or other adverse medical event the appeared for the first time or worsened during participation in the study AND were associated with the intervention in the study - urine collection. Serious adverse events were study defined adverse events that were considered life-threatening.
  Only events considered associated with the intervention in the study - urine collection- were collected.
Arm/Group | NINJA
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

LIMITATIONS AND CAVEATS:
This study had a relatively small sample size with only 27 participants developing AKI. Additionally, this study was performed in non-critically ill children and the findings may not be applicable to a broader population of hospitalized children and adults.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03527160/Prot_SAP_000.pdf